CLINICAL TRIAL: NCT04335799
Title: Improving Weight Loss Outcomes of Black Women Using a Culturally-Relevant Stress-Management Enhanced Behavioral Weight Loss Intervention
Brief Title: Reducing Weight and Elevated Stress Levels Using Educational and Behavioral Tools
Acronym: RESET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: MCC-21236; R01DK125367 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-04-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Loss Plus Stress Management (Experimental): Diabetes Prevention Program Intensive Lifestyle Intervention augmented with stress management training
  Interventions: Behavioral: Diabetes Prevention Program Intensive Lifestyle Intervention plus stress management training
- Weight Loss Only (Active Comparator): Diabetes Prevention Program Intensive Lifestyle Intervention plus general women's health topics
  Interventions: Behavioral: Diabetes Prevention Program Intensive Lifestyle Intervention plus general women's health topics

INTERVENTIONS:
Behavioral: Diabetes Prevention Program Intensive Lifestyle Intervention plus stress management training — 12-month evidence based weight loss intervention with additional training on stress management strategies
  Arms: Weight Loss Plus Stress Management
Behavioral: Diabetes Prevention Program Intensive Lifestyle Intervention plus general women's health topics — 12-month evidence based weight loss intervention with an attention control of general women's health topics
  Arms: Weight Loss Only

SUMMARY:
The purpose of this protocol is to test the effects on weight of an evidence-based behavioral weight loss program enhanced with culturally targeted stress management strategies compared to the evidence-based weight loss program alone among adult black females with obesity and elevated stress levels. Participants will be randomized to receive either a behavioral weight loss intervention with a focus on stress management or the weight loss intervention alone for 26 sessions.

ELIGIBILITY:
Inclusion Criteria:

* BMI of at least 30 kg/m^2
* elevated stress levels based on perceived stress scale score
* self-identified as black race

Exclusion Criteria:

* pregnant or are planning to become pregnant in the next year
* known major medical or psychological condition known to influence body weight loss (e.g., medicated or poorly controlled diabetes (fasting blood glucose > 126 mg/dL), cardiovascular event in the preceding 12 months, history of gastric bypass surgery, bariatric surgery, or eating disorder)
* history of psychiatric hospitalization in past 2 years
* history of substance abuse or eating disorder
* any condition for which a medical professional has suggested diet modification, physical activity, and/or weight reduction would be contraindicated.
* currently taking medications for weight loss

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
4-month mean weight change of participants using SECA scale | Baseline to Month 4
  weight change as measured by a SECA scale in kilograms and baseline and month 4 will be calculated and averaged
12-month mean weight change of participants using SECA scale | Baseline to Month 12
  weight change as measure by a SECA scale in kilograms and baseline and month 12 will be calculated and averaged

SECONDARY OUTCOMES:
mean change in perceived stress using Perceived Stress Scale-10 score | Baseline to Month 4
  Perceived stress as measured with a validated survey will be assessed at baseline and month to assess changes in participant's stress
mean change in perceived stress using Perceived Stress Scale-10 score | Baseline to Month 12
  Perceived stress as measured with a validated survey will be assessed at baseline and month 12 to assess changes in participant's stress

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Carson, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buro AW, Baskin M, Miller D, Ward T, West DS, Gore LR, Gwede CK, Epel E, Carson TL. Rationale and study protocol for a randomized controlled trial to determine the effectiveness of a culturally relevant, stress management enhanced behavioral weight loss intervention on weight loss outcomes of black women. BMC Public Health. 2022 Jan 28;22(1):193. doi: 10.1186/s12889-022-12519-z. PMID 35090433
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinicaltrialssearch/?diseasesite=&query=21236&studytype=&medication=&therapy=&pi=&nct=&sortcriteria=